CLINICAL TRIAL: NCT01464138
Title: Evaluation of Fosmidomycin and Clindamycin in the Treatment of Acute Uncomplicated Plasmodium Falciparum Malaria in Children
Brief Title: Evaluation of Fosmidomycin and Clindamycin in the Treatment of Acute Uncomplicated P.Falciparum Malaria in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jomaa Pharma GmbH (Industry)
Collaborators: Fundacio Clinic Barcelona (Other); Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JP012
Record Dates: First submitted 2009-10-26; First posted 2011-11-03 (Estimated); Last update posted 2011-11-03 (Estimated); Status verified 2011-11

CONDITIONS: Malaria
Keywords: Malaria
MeSH Terms: conditions — Malaria | interventions — fosmidomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fosmidomycin-Clindamycin (Experimental): Single arm study. Co-administration of Fosmidomycin and Clindamycin.
  Interventions: Drug: Fosmidomycin and Clindamycin co-administration

INTERVENTIONS:
Drug: Fosmidomycin and Clindamycin co-administration — Fosmidomycin sodium syrup at a concentration of 250mg/5ml and clindamycin hydrochloride syrup at a concentration of 75mg/5ml. Administered in doses of fosmidomycin 30mg/kg/dose + clindamycin 10mg/kg/dose twice daily for three days (total daily dose fosmidomycin 60mg/kg, clindamycin 20mg/kg)

SUMMARY:
This is an open label uncontrolled study to determine the efficacy of fosmidomycin and clindamycin when co-administered orally over three days in the treatment of acute uncomplicated Plasmodium falciparum malaria in children.

The primary study endpoints will be the cure rate on Day 28 (PCR corrected). The secondary endpoints will be the cure rate on Day 7 and the parasite and fever clearance times.

DETAILED DESCRIPTION:
An open label uncontrolled study to determine the efficacy of fosmidomycin and clindamycin when co-administered orally over three days in the treatment of acute uncomplicated Plasmodium falciparum malaria in children.

The primary study endpoints will be the cure rate on Day 28 (PCR corrected). The secondary endpoints will be the cure rate on Day 7 and the parasite and fever clearance times.

Study population A total of 40 children will be recruited into the study. Sample size calculations have been made on the basis that this trial aims at substantiating the efficacy results obtained in children in Gabon. In the largest trial of this drug combination done in Gabon, 51 children were recruited, and the per-protocol, PCR-adjusted day 28 cure rate was 89% (42/47; 95% CI, 77 to 96%). Based on this expected 90% efficacy estimate, a sample size of 35 children produces a two-sided 95% confidence interval with a an estimated precision of 20%.

Allowing for an attrition rate of 10% for non-evaluable subjects, a sample size of 40 subjects will be required.

Study endpoints Primary The primary endpoint will be the cure rate on Day 28 (PCR corrected). Secondary The secondary endpoints will be the cure rate on Day 7 and the parasite and fever clearance times.

Withdrawal criteria during treatment (classified as therapeutic failure)

* Severe deterioration in clinical condition
* Signs of severe malaria, according to WHO criteria
* Onset of drug related serious adverse events
* Repeated vomiting within one hour of re-dosing

Discontinuation criteria after completion of treatment (classified as therapeutic failure)

* Persistent parasitaemia at 96 hours after initiation of treatment
* Parasitaemia during follow-up period after initial clearance
* No reduction of parasitaemia within 48 hours after initiation of treatment
* Onset of drug related serious adverse events

Discontinuation criteria after completion of treatment (not classified as therapeutic failure)

* Withdrawal of guardian consent
* Loss to follow up
* Protocol violation Procedure for treatment The study drugs will be administered under direct supervision by a study clinician or nurse in doses of fosmidomycin 30mg/kg/dose + clindamycin 10mg/kg/dose twice daily for three days (total daily dose fosmidomycin 60mg/kg, clindamycin 20mg/kg).

In the event of vomiting within one hour of dosing, the same dose of each drug will be re-administered from a supplemental drug supply.

Re-dosing will be done only once for each drug administration and only twice for the whole of the treatment period.

Concomitant treatment Subjects will be treated for symptoms and adverse events during the study period by standard treatment.

Drugs with antimalarial activity or likely to have an effect on parasitaemia will not be permitted during the study. This will include artemether-lumefantrine combination, artesunate, sulfadoxine/pyrimethamine combination, chloroquine, amodiaquine and co-trimoxazole.

Trial procedures and duration of the study A general physical examination will be performed on admission to the study. All subjects will be hospitalised for a minimum of three days until they are asymptomatic and aparasitaemic.

Brief examinations will be conducted daily during this period and once weekly thereafter to assess general physical status.

Thereafter subjects will return for out-patient follow-up on days 7 ± 1 day, 14 ± 2 days, 21 ± 2 days and 28 ± 2 days.

All subjects are expected to participate in the trial for the total duration of 28 days.

Those subjects not attending for follow-up will be located by a member of the study staff who will provide transportation to the hospital for the scheduled examinations or ascertain the reason for failing to attend.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged six months to three years
* Female subjects aged six months to three years
* Body weight >5kg
* Acute (symptoms lasting less than 14 days) uncomplicated P falciparum malaria
* Asexual parasitaemia between 1,000/µL and 200,000/µL
* Ability to tolerate oral therapy
* Willingness of the parent or guardian to provide informed signed consent

Exclusion Criteria:

* Symptoms/signs of severe malaria, according to WHO criteria
* Body weight <5kg
* Other plasmodial infections (P vivax, P ovale, P malariae)
* Severe malnutrition with weight for age <60% or clinical kwashiorkor
* Gastro-intestinal disturbance with persistent vomiting (> three episodes within previous 24 hours) and/or diarrhoea (> 5 loose stools in the preceding 24 hours)
* Concomitant disease masking assessment of response including sickle cell disease and severe cardiac, hepatic or renal impairment
* Haemoglobin <7g/dl
* Adequate anti-malarial treatment within previous 7 days
* Inability to tolerate oral therapy
* Parent or guardian deemed to be unsupportive
* On co-trimoxazole prophylaxis

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Day 28 cure rate >95% | 28 days

SECONDARY OUTCOMES:
Day 7 cure rate of 100% | Day 6
Parasite Clearance Time | 0-7 days
Fever Clearance Time | 0-7 days

CONTACTS AND LOCATIONS:
Overall Officials: Quique Bassat, PhD, Principal Investigator — CRESIB, Barcelona
Locations (1):
- Centro de Investigacao em Saude da Manhica, Maputo, Mozambique